CLINICAL TRIAL: NCT04107168
Title: An Observational Study to Evaluate the Microbiome as a Biomarker of Efficacy and Toxicity in Cancer Patients Receiving Immune Checkpoint Inhibitor Therapy
Brief Title: Microbiome Immunotherapy Toxicity and Response Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Microbiotica Ltd (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Pippa Corrie, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: MITRE; C7535/A27717 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2019-09-09; First posted 2019-09-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Melanoma; Renal Cancer; Lung Cancer
Keywords: NSCLC; Advanced; Unresectable; Microbiome; Adjuvant; Resected; Immune checkpoint inhibitors
MeSH Terms: conditions — Melanoma; Kidney Neoplasms; Lung Neoplasms | interventions — Nivolumab; pembrolizumab; Ipilimumab; durvalumab; tremelimumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research blood samples, saliva samples and stool samples collected. Tumour samples and organ sample after toxicity if available. A single, optional nasopharyngeal swab for COVID-19 may be offered to participants before study entry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Cohort 1: Disease: Unresectable AJCC (American Joint Committee on Cancer) stage 3 or 4 melanoma.
  Anti-PD-1 monotherapy (Nivolumab or Pembrolizumab). Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab
- Cohort 2: Disease: Unresectable AJCC stage 3 or 4 melanoma. Nivolumab + Ipilimumab. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Cohort 3: Disease: Advanced renal cell carcinoma. Anti-PD-(L)1 + kinase inhibitor. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab
- Cohort 4: Disease: Advanced renal cell carcinoma Nivolumab + Ipilimumab. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Cohort 5: Disease: Advanced NSCLC Anti-PD-(L)1 (Nivolumab, Pembrolizumab or Atezolizumab) monotherapy in the first line setting. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Drug: Atezolizumab
- Cohort 6: Disease: Advanced NSCLC Anti-PD-(L)1 (Nivolumab, Pembrolizumab or Atezolizumab) + chemotherapy +/- antiangiogenic (Bevacizumab) in the first line setting. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Bevacizumab
- Cohort 7: Disease: Resected AJCC stage 3 or 4 melanoma. Anti-PD-1 monotherapy (Nivolumab or Pembrolizumab). Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab
- Cohort 8: Disease: Resected renal cancer Anti-PD-(L)1 monotherapy (Durvalumab or Pembrolizumab). Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Pembrolizumab; Drug: Durvalumab
- Cohort 9: Disease: Resected renal cancer Durvalumab + Tremelimumab. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Nivolumab — A human immunoglobulin G4 (IgG4) monoclonal antibody, which binds to the programmed death-1 receptor (PD-1).
  Other Names: Opdivo
  Groups: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7
Drug: Pembrolizumab — A human immunoglobulin G4-kappa (IgG4-kappa) monoclonal antibody that targets PD-1.
  Other Names: Keytruda
  Groups: Cohort 1; Cohort 5; Cohort 6; Cohort 7; Cohort 8
Drug: Ipilimumab — A human immunoglobulin G1 (IgG1) monoclonal antibody raised against cytotoxic T lymphocyte antigen-4 (CTLA-4).
  Other Names: Yervoy
  Groups: Cohort 2; Cohort 4
Drug: Durvalumab — A human immunoglobulin G1-kappa (IgG1-kappa) monoclonal antibody that binds to programmed death ligand 1 (PD-L1).
  Other Names: Imfinzi
  Groups: Cohort 8; Cohort 9
Drug: Tremelimumab — A fully human monoclonal antibody raised to target cytotoxic T lymphocyte-associated antigen 4 (CTLA-4).
  Other Names: CP-675,206
  Groups: Cohort 9
Drug: Atezolizumab — A humanised IgG1 monoclonal antibody raised to target programmed death-ligand 1 (PD-L1).
  Other Names: Tecentriq
  Groups: Cohort 5; Cohort 6
Drug: Bevacizumab — A humanised IgG1 monoclonal antibody raised to target vascular endothelial growth factor (VEGF).
  Other Names: Avastin
  Groups: Cohort 6

SUMMARY:
This is a observational study to investigate how the microbiome correlates with efficacy and toxicity of immune checkpoint inhibitors in patients with advanced cancer.

DETAILED DESCRIPTION:
The gastrointestinal microbiome of a healthy individual is comprised of many hundreds of bacteria species and thousands of bacteria strains. The composition of bacteria in an individual's microbiome can change over time and this can be influenced by factors including diet, drugs, genetics and infection. These bacteria play a central role in digestion of food, development and regulation of our immune system as well as our resistance to pathogens. Recent evidence suggest that a patient's intestinal microbiota composition plays a critical, though as yet poorly defined, role in determining both therapeutic efficacy and likelihood of significant adverse events to T-cell checkpoint inhibitor immunotherapy.

Immune checkpoint inhibitors are revolutionising treatment of many types of metastatic cancer, including melanoma, renal and non-small cell lung cancer, in the expectation of improving patient overall survival. However, they have limitations as they do not work for all patients and can cause unpredictable, complex immune-related toxicities. The investigators will perform a detailed study of cancer patients receiving checkpoint inhibitors. Saliva and a series of stool samples will be collected from each patient to analyse their microbiome and will be linked to treatment response, by examining blood samples and - if available - tumour and organ samples. The investigators hope this work will enable personalisation of patient immunotherapies based on microbiome biomarkers, as well as precisely manipulate a patient's microbiota to optimise their immunotherapy.

In addition, participants who have consented to take part in an optional sub-study may be offered a single nasopharyngeal swab for COVID-19 antigen before study entry. The investigators hope that that this identify correlations between the microbiome and COVID-19.

Comparison with a limited cohort of healthy household members (up to 360 volunteers) acting as controls will provide additional essential information about the role of the patient-specific microbiome.

ELIGIBILITY:
Inclusion Criteria for cancer patients:

* Signed informed consent

  * Aged ≥18 years old
  * Histological or cytological confirmation of invasive malignancy
  * Due to commence palliative, adjuvant or neoadjuvant systemic therapy including an anti-PD-(L)1 antibody +/- anti-CTLA-4 antibody
  * Patients with unresectable disease must have radiologically and/or clinically measurable disease, by RECIST version 1.1; target lesions must not have been previously irradiated; baseline tumour assessments must be performed within 45 days prior to starting immune checkpoint inhibitor treatment
  * Received no prior immune checkpoint inhibitors (previous treatment with other types of anti-cancer therapy is determined by patient cohort; for patients with unresectable disease, prior adjuvant therapy with immune checkpoint inhibitor(s) is allowed).
  * Willing and able to comply with scheduled visits, treatment plans, sample collections and other study procedures

Exclusion Criteria for cancer patients:

* Other invasive malignancies diagnosed within the last year which are not fully resected, or in complete remission, or for which additional therapy is required
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the investigator would place the patient at undue risk, or interfere with their ability to comply with the study. Examples may include, but are not limited to:

  * Patients with uncontrolled ischaemic heart or other cardiovascular event (e.g. myocardial infarction, new angina, stroke, transient ischaemic attack, or new congestive cardiac failure) within the last 6 months
  * Presence of active infection
  * Cirrhotic liver disease, known chronic active or acute hepatitis B, or hepatitis C
  * Current active, severe, or uncontrolled autoimmune condition, including but not limited to Crohn's disease and ulcerative colitis.
* Women who are pregnant, plan to become pregnant or are lactating during the study period.
* Requirement for non-physiological dose of oral steroids, or regular use of any other immunosuppressive agents; less than 10mg prednisolone or equivalent doses are allowed. Use of inhaled or topical steroids is allowed.

Household control eligibility requirements:

Confirmation of suitability to be a household control participant will be determined by completing a self-assessed questionnaire either at home or in clinic.

Household controls must:

* NOT have had any gastrointestinal infections i.e., parasites, viruses or diarrhoeal episodes during the last 6 months.
* NOT have taken antibiotics for at least 6 months
* NOT have or be recovering from any chronic intestinal disease such as:

  * Crohn's disease
  * Ulcerative colitis
  * Coeliac disease
  * Irritable bowel syndrome
  * Stomach ulcers
* NOT have a chronic autoimmune disease or significant allergies e.g., multiple sclerosis, asthma requiring regular medication, psoriasis.
* NOT have and NOT be recovering from any form of cancer.
* NOT take proton pump inhibitors, steroids, other non-steroidal anti-inflammatory drugs such as ibuprofen or aspirin.
* NOT had requirement to be hospitalised for treatment of COVID-19

In addition, household controls must sign informed consent and be aged ≥18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 1800 cancer patients due to receive anti-PD(L)1 +/- anti-CTLA-4 antibodies for treatment of their cancer and up to 360 consenting adults (household controls) who live with one of these cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-07-08 (Estimated); Study Completion 2025-07-08 (Estimated)

PRIMARY OUTCOMES:
Can the microbiome signature predict progression-free survival (PFS) of 1 year or greater | Minimum 1 year PFS
  The primary outcome measure is the ability to predict for PFS of 1 year or greater for patients with advanced melanoma, renal and non-small cell lung cancer (cohorts 1-6).

SECONDARY OUTCOMES:
Can the microbiome signature predict PFS | 1 year & 2 years PFS
  Measure the ability of the microbiome signature to predict 6 month PFS, 2 year PFS, overall response rate and median PFS in Cohorts 1-6.
Can the microbiome signature overall survival (OS) | Up to 6 years
  Measure the ability of the microbiome signature to median OS in Cohorts 1-6.
Can the microbiome signature to predict relapse | 1 year & 2 years relapse-free survival (RFS)
  Measure the ability of the microbiome signature to predict for 1 or 2 year relapse after resection of high risk melanoma or renal cancer in cohorts 7-9.
Does the microbiome correlate with treatment efficacy | Up to 6 years
  To compare pre-treatment oral and gut microbiome findings and their association with treatment efficacy.
Correlate microbiome findings with incidence and characteristics of immune-related adverse events | Up to 6 years
  To correlate microbiome findings with incidence and characteristics of CTCAE V5-defined Grade 3 or greater immune-related adverse events in all enrolled cancer patients, and any association with response to immunosuppressants.
Correlation microbiome findings and known characteristics of patients | Up to 6 years
  To correlate microbiome findings with aspects of pre-existing patient characteristics and behaviour including but not limited to diet, smoking history, BMI, use of antibiotics, steroids, proton pump inhibitors, non-steroidal anti-inflammatory drugs and probiotics.
Control for the microbiome of cancer patients | Up to 6 years
  To compare the microbiome signature of cancer patients with a household control group of people who are not known to have cancer.
Build a library of biological samples for future research | Up to 6 years
  To retain a library of biological samples (saliva, stool, blood and tumour as well as organ if available) with linked patient data for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, Principal Investigator — Cambridge University Hospital
Locations (13):
- United Kingdom (13):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - University Hospitals Dorest NHS Foundation Trust, Bournemouth
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre University NHS Trust, Cardiff
  - Western General Hospital, Edinburgh
  - The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust, Kings Lynn
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Somerset NHS Foundation Trust, Taunton
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson NA, Stewart GD, Welsh SJ, Doherty GJ, Robinson MJ, Neville BA, Vervier K, Harris SR, Adams DJ, Dalchau K, Bruce D, Demiris N, Lawley TD, Corrie PG. The MITRE trial protocol: a study to evaluate the microbiome as a biomarker of efficacy and toxicity in cancer patients receiving immune checkpoint inhibitor therapy. BMC Cancer. 2022 Jan 24;22(1):99. doi: 10.1186/s12885-021-09156-x. PMID 35073853